CLINICAL TRIAL: NCT04216264
Title: Pilot Adaptive Tool To Encourage Risk Reduction in iNfancy (PATTERN)
Brief Title: Pattern - Reach Aim 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Pro00102738; U54MD012530 (NIH)
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Results first posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-10

CONDITIONS: Obesity
Keywords: infant; mother-baby
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Response (Other)
  Interventions: Behavioral: Standard response
- Non-response (Other)
  Interventions: Behavioral: Targeted response

INTERVENTIONS:
Behavioral: Standard response — Parents pick from a menu of behavior changes
  Arms: Response
Behavioral: Targeted response — Stepped up phone interaction with parents based on menu of behavior changes
  Arms: Non-response

SUMMARY:
The purpose of this research study is to learn about different approaches to promoting healthy growth among infants, and understanding parents' likes and dislikes of an approach to reducing risk factors for obesity later in life. The study includes filling out some forms with questions about your baby and your thoughts about your baby's growth and health, and engaging in a pattern of changes in or prevention of risk factors in the first year of life. Parents will receive information about changes and some tools and materials to take home with them. Some parents may receive phone calls between visits as well. The study takes place from soon after birth through the infant's age of 9 months. The estimated total time of interaction between the study staff and parents during the study period is 4 hours.

DETAILED DESCRIPTION:
As this is a dyad study, each dyad is considered to be a participant and demographic information will reflect the infant in the dyad, per parent report.

ELIGIBILITY:
Inclusion Criteria:

* Non-Hispanic black (as documented in MaestroCare) parents/caregivers with; infants ages 2 weeks to 2 months of age; infant birthweight between 2500g and 4000g; infant gestational age is at least 36 weeks

Exclusion Criteria:

* non-English-speaking; infant with serious disease or disorder affecting growth and nutrition

Ages: 2 Weeks to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2020-05-07 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Wood, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants are recruited as caregiver/child dyads.
Pre-assignment Details: Participants will be screened for eligibility and if eligible and they consent, complete a questionnaire identifying current potential risks for obesity in infancy. Once one of the three domains is identified, parents will be given scripted educational and supportive messaging relevant to the domain.
Groups:
- Standard Response Caregiver/Child Dyad - Caregiver; Standard Response Caregiver/Child Dyad - Child: Standard response: Parents pick from a menu of behavior changes
- Targeted Response Caregiver/Child Dyad - Caregiver; Targeted Response Caregiver/Child Dyad - Child: Targeted response: Stepped up phone interaction with parents based on menu of behavior changes
Period: Overall Study
Arm/Group | Standard Response Caregiver/Child Dyad - Caregiver | Standard Response Caregiver/Child Dyad - Child | Targeted Response Caregiver/Child Dyad - Caregiver | Targeted Response Caregiver/Child Dyad - Child
Started | 7 | 7 | 7 | 7
Completed | 5 | 5 | 2 | 2
Not Completed | 2 | 2 | 5 | 5

BASELINE CHARACTERISTICS:
Population: Demographic information was not collected on parents/caregivers. The unit of analysis was the dyad, with demographic information reflecting the parent-reported demographics of their infant only.
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Response Caregiver/Child Dyad - Child | Targeted Response Caregiver/Child Dyad - Child | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 7 | 14
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 1 (1.1) | 1 (1.3) | 1 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Satisfied or Very Satisfied With Information Given to Them, as Measured by Follow up Questionnaire
Description: Completed Likert scale with 1=very unsatisfied, 2=unsatisfied, 3=neutral, 4=satisfied, 5=very satisfied
Time Frame: 3 to 6 months after baseline assessment
Population: Caregiver/child dyads who completed the study.
Measure: Count of Participants; unit: Participants
Groups:
- Standard Response Caregiver/Child Dyads: Standard response: Parents pick from a menu of behavior changes
- Targeted Response Caregiver/Child Dyads: Targeted response: Stepped up phone interaction with parents based on menu of behavior changes
Arm/Group | Standard Response Caregiver/Child Dyads | Targeted Response Caregiver/Child Dyads
Number analyzed (Participants) | 5 | 2
Participants | 4 | 2

2. Primary Outcome: Percentage of Successful Contacts With Families Via Telephone and/or in Clinic
Description: Number of successful contacts with families divided by number of attempts to contact by research staff x 100
Time Frame: 3 to 6 months after baseline assessment
Population: Participants with data collected.
Measure: Number; unit: percentage of contacts
Arm/Group | Standard Response Caregiver/Child Dyads | Targeted Response Caregiver/Child Dyads
Number analyzed (Participants) | 7 | 3
percentage of contacts | 85.8 | 100

3. Secondary Outcome: Percent of Participants Exclusively Breastfeeding at 4 Months Postnatal Age
Description: Dyad caregivers were asked what type of milk was being consumed by the infant, with 4 options available: 1) Formula only, 2) Mostly formula and some breast milk, 3) Mostly breast milk, but some formula, or 4) Breast milk only.
Time Frame: 3 to 6 months after baseline assessment
Population: Participants with data collected.
Measure: Number; unit: percentage of participants
Arm/Group | Standard Response Caregiver/Child Dyads | Targeted Response Caregiver/Child Dyads
Number analyzed (Participants) | 7 | 3
percentage of participants | 71.4 | 33.3

4. Secondary Outcome: Percent of Participants Delaying Complementary Feeding Until 4 Months Postnatal Age
Description: Dyads caregivers were asked, "Is your baby eating solid foods yet or do you put any solid foods in the bottle?", with 2 options available: 1) Yes or 2) No
Time Frame: 3 to 6 months after baseline assessment
Population: Participants with data collected.
Measure: Number; unit: percentage of participants
Arm/Group | Standard Response Caregiver/Child Dyads | Targeted Response Caregiver/Child Dyads
Number analyzed (Participants) | 7 | 3
percentage of participants | 71.4 | 33.3

5. Secondary Outcome: Percent of Participants Reporting "Never" Engaging in Screentime While Feeding and With '0' Minutes of Active TV Watching at 4 Months Postnatal Age
Description: Dyad caregivers were asked "I watch TV or look at or use my phone while feeding my baby" and responded with one of 5 Likert-scale responses: 1) Never, 2) Seldom, 3) Half of the time, 4) Most of the time, 5) Always
Time Frame: 3 to 6 months after baseline assessment
Population: Participants with data collected.
Measure: Number; unit: percentage of participants
Arm/Group | Standard Response Caregiver/Child Dyads | Targeted Response Caregiver/Child Dyads
Number analyzed (Participants) | 7 | 3
percentage of participants | 42.9 | 100

ADVERSE EVENTS:
Time Frame: Approximately 7 months
Description: Participants are treated as dyad, but adverse events refer to infant only. Adverse events were not collected for caregivers.
Groups:
- Standard Response Caregiver/Child Dyad - Child: Standard response: Dyads pick from a menu of behavior changes
- Targeted Response Caregiver/Child Dyad - Child: Targeted response: Stepped up phone interaction with dyads based on menu of behavior changes
Arm/Group | Standard Response Caregiver/Child Dyad - Child | Targeted Response Caregiver/Child Dyad - Child
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/64/NCT04216264/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/64/NCT04216264/ICF_001.pdf